CLINICAL TRIAL: NCT03196622
Title: Validation of a Screening Test of Sarcopenia in the Elderly People at Hospital and in Retirement Houses
Brief Title: Validation of a Screening Test for Sarcopenia in Older People
Acronym: SARCSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Nutriset (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHU-339; 2016-A01254-47 (Other: 2016-A01254-47)
Record Dates: First submitted 2017-06-21; First posted 2017-06-23 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Elderly people; Hospitalization
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Masking Description: Open
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Older people (Experimental): A cross-sectional multicentre study will be performed in hospital and retirement houses on patients ages 75 years old or more.
  Interventions: Device: Handgrip test

INTERVENTIONS:
Device: Handgrip test — Handgrip strenght can be used in daily clinical practice to screen patients having sarcopenia to improve treatment and quality of life.

SUMMARY:
Identify the threshold which the handgrip strenght can be used as a screening test of sarcopenia.

Handgrip strenght can be used in daily clinical practice to screen patients having sarcopenia to improve treatment and quality of life.

DETAILED DESCRIPTION:
A cross-sectional multicentre study will be performed in hospital and retirement houses on patients ages 75 years old or more.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 75 years old

Exclusion Criteria:

* Palliative care,
* Protection of vulnerable adults

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2017-07-11 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Handgrip test could be used as a screening test of sarcopenia | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Marie BLANQUET, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France